CLINICAL TRIAL: NCT02528903
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single-ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of MHAB5553A in Healthy Volunteers
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of MHAB5553A in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: GV29827
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — lesofavumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Cohort A (Experimental)
  Interventions: Drug: MHAB5553A; Drug: Matching placebo
- Cohort B (Experimental)
  Interventions: Drug: MHAB5553A; Drug: Matching placebo
- Cohort C (Experimental)
  Interventions: Drug: MHAB5553A; Drug: Matching placebo
- Cohort D (Experimental)
  Interventions: Drug: MHAB5553A; Drug: Matching placebo
- Cohort E (Experimental)
  Interventions: Drug: MHAB5553A; Drug: Matching placebo

INTERVENTIONS:
Drug: MHAB5553A — Single intravenous administration, at various doses, depending on the cohort
Drug: Matching placebo — Single intravenous dose

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single-ascending dose study in healthy volunteers to investigate the safety, tolerability, and pharmacokinetics (PK) of MHAB5553A.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF)
* Body mass index (BMI) between 18 and 32 kg/m2, inclusive
* Weight 40-100 kg
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, and vital signs
* Clinical laboratory evaluations should be within reference range for the test, unless deemed not clinically significant by the investigator and sponsor at screening
* Willing to abstain from using drugs of abuse while enrolled in the study
* Willing and able to comply with protocol-specified criteria in regard to contraceptive protection
* Able to comply with the study protocol, in the investigator's judgment

Exclusion Criteria:

* History or clinically significant manifestations of metabolic, hepatic, renal, hematologic, immunodeficiency, pulmonary, cardiovascular, gastrointestinal, urologic, neurologic, or psychiatric disorders
* History of anaphylaxis, hypersensitivity or drug allergies, unless approved by the investigator and sponsor
* History or presence of an abnormal ECG, which, in the investigator's or sponsor's opinion, is clinically significant (including evidence of previous acute myocardial infarction, complete left bundle branch block, second-degree heart block, or complete heart block)
* History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit
* History of significant drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to screening visit or hard drugs (such as cocaine, phencyclidine [PCP], and crack) within 1 year prior to screening
* Current tobacco smokers (positive history within 3 months before initiation of dosing on Day 1), or those with positive cotinine test at check-in
* Positive drug screen at screening or at check-in
* Positive pregnancy test result at screening or Day -1 or breast feeding during the study
* Any serious medical condition or abnormality in clinical laboratory tests that, in the investigator's judgment, precludes the participant's safe enrollment in and completion of the study
* Unwillingness to comply or other conditions that, in the opinion of the investigator, would interfere with the ability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2016-01-26 (Actual); Study Completion 2016-01-26 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events, graded by severity | Until study discontinuation/termination, up to 120 days
Changes in vital signs during and following MHAB5553A administration | Throughout the study, up to 120 days
Changes in physical examination finding during and following MHAB5553A administration | Throughout the study, up to 120 days
Changes in clinical laboratory results during and following MHAB5553A administration | Throughout the study, up to 120 days
Changes in electrocardiogram (ECG) findings during and following MHAB5553A | Throughout the study, up to 120 days
Incidence of serum anti-MHAB5553A antibodies | Until study discontinuation/termination, up to 120 days

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of MHAB5553A | Up to 120 days
Time to Cmax (tmax) of MHAB5553A | Up to 120 days
Area under the concentration-time curve up to last measurable time point (AUC0-last) of MHAB5553A | Up to 120 days
Area under the concentration-time curve extrapolated to infinity (AUC0-inf) of MHAB5553A | Up to 120 days
Clearance (CL) of MHAB5553A | Up to 120 days
Volume of distribution at steady-state (Vss) of MHAB5553A | Up to 120 days
Terminal elimination half-life (t1/2) of MHAB5553A | Up to 120 days
Mean Residence Time (MRT) of MHAB5553A | Up to 120 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- inVentiv Health Clinique, Québec, Canada

REFERENCES:
- [Derived] Lim JJ, Derby MA, Zhang Y, Deng R, Larouche R, Anderson M, Maia M, Carrier S, Pelletier I, Girard J, Kulkarni P, Newton E, Tavel JA. A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending-Dose Study To Investigate the Safety, Tolerability, and Pharmacokinetics of an Anti-Influenza B Virus Monoclonal Antibody, MHAB5553A, in Healthy Volunteers. Antimicrob Agents Chemother. 2017 Jul 25;61(8):e00279-17. doi: 10.1128/AAC.00279-17. Print 2017 Aug. PMID 28559255